CLINICAL TRIAL: NCT06500286
Title: Comparison Between Dorsal Nerve Block and Caudal Block Effect in Post Operative Pain in Hypospedius Repair in Children
Brief Title: Dorsal Nerve Block and Caudal Block in Hypospedius Repair in Children
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Soha Abd Elhamid Fawzy, Resident doctor in assiut university hospitals, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dorsal block in hypospedius
Record Dates: First submitted 2024-03-10; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Dorsal Nerve Block in Hypospiudus
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): • Group A receive caudal block placing the patient into the left lateral decubitus position. . The sacral hiatus was found by palpating the sacral cornu and a 22-G needle was placed through it. After passing through the sacrococcygeal 0.25% bupivacaine was administered at a dose of 0.2 ml/kg.the procedure was completed, the patient was placed into the supine Position.
  Interventions: Drug: Marciane
- Group B (Experimental): Group B US guided Dorsal penil block. The 5-10 MHz linear probe was placed at the penis root, making it possible to observe the corpus cavernosum, corpus spongiosum, dorsal artery and vein, and the deep penile fascia (Buck's fascia) on the transverse plane with gentle penile traction. The in-plane technique was then used to insert a 50-mm block needle toward the dorsal penile section from the lateral part of the penis root. The needle was then advanced from the hyperechoic superficial penis fascia (Dartos fascia) and the superficial sheath was passed. After advancing the needle into Buck's fascia, the needle was placed lateral to the dorsal artery, at a position between Buck's fascia and tunica albuginea. Negative aspiration was performed. US was then used to observe the distribution of the anesthetic while half of the total 0.25% bupivacaine dose (0.2 mL/kg) was administered (Fig. 1). Afterward, the same procedure was also performed on the other side of the penis.
  Interventions: Drug: Marcaine

INTERVENTIONS:
Drug: Marciane — Group A caudal block 0.25% bupivacaine was administered at a dose of 0.2 ml/k
  Other Names: bupivacaine
  Arms: Group A
Drug: Marcaine — Dorsal penil block 0.25% bupivacaine was administered at a dose of 0.2 ml/k
  Other Names: bupivacaine
  Arms: Group B

SUMMARY:
Comparison between Dorsal nerve block and caudal block effect in post operative pain in hypospedius repair in children Randomoized clinical trial

DETAILED DESCRIPTION:
• Group A receive caudal block placing the patient into the left lateral decubitus position. Povidone iodine was used to sterilize the skin. The sacral hiatus was found by palpating the sacral cornu and a 22-G needle was placed through it. After passing through the sacrococcygeal membrane by using the loss of resistance method, the caudal epidural space was entered. Negative aspiration was used to make sure there was no blood or cerebrospinal fluid present and 0.25% bupivacaine was administered at a dose of 0.2 ml/kg. Once the procedure was completed, the patient was placed into the supine Position.

Group B US guided Dorsal penil block. General anesthesia induction was followed by skin sterilization using 70% alcohol in 2% chlorhexidine. The 5-10 MHz linear probe was placed at the penis root, making it possible to observe the corpus cavernosum, corpus spongiosum, dorsal artery and vein, and the deep penile fascia (Buck's fascia) on the transverse plane with gentle penile traction. The in-plane technique was then used to insert a 50-mm block needle toward the dorsal penile section from the lateral part of the penis root. The needle was then advanced from the hyperechoic superficial penis fascia (Dartos fascia) and the superficial sheath was passed. After advancing the needle into Buck's fascia, the needle was placed lateral to the dorsal artery, at a position between Buck's fascia and tunica albuginea. Negative aspiration was performed. US was then used to observe the distribution of the anesthetic while half of the total 0.25% bupivacaine dose (0.2 mL/kg) was administered (Fig. 1). Afterward, the same procedure was also performed on the other side of the penis.

ELIGIBILITY:
Inclusion Criteria:

* aged 2-12 years
* ASA physical status I or II

Exclusion Criteria:

* asthmatic patients
* emergency surgery
* intellectual disability
* neurological diseases with agitation-like symptoms
* renal or hepatic disease,
* cardiac or respiratory disease
* allergy to the study drugs
* parent refusal
* psychiatric diseases

Ages: 2 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 103 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of dorsal penile block | 1year
  Score of pain visual Analougue Score

SECONDARY OUTCOMES:
Comparison between post operative analegesia effect and side effect of dorsal penileblock and caudal block | 1year
  Comparison between post operative analegesia effect and side effect of dorsal penileblock and caudal block

CONTACTS AND LOCATIONS:
Overall Officials: Soha Abdelhamid Fawzy, Resident, Principal Investigator — Resident

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baskin LS, Lee YT, Cunha GR. Neuroanatomical ontogeny of the human fetal penis. Br J Urol. 1997 Apr;79(4):628-40. doi: 10.1046/j.1464-410x.1997.00119.x. PMID 9126098
- [Result] Ngoo A, Borzi P, McBride CA, Patel B. Penile nerve block predicts higher revision surgery rate following distal hypospadias repair when compared with caudal epidural block: A consecutive cohort study. J Pediatr Urol. 2020 Aug;16(4):439.e1-439.e6. doi: 10.1016/j.jpurol.2020.05.150. Epub 2020 Jun 6. PMID 32636118
- [Result] Hueber PA, Salgado Diaz M, Chaussy Y, Franc-Guimond J, Barrieras D, Houle AM. Long-term functional outcomes after penoscrotal hypospadias repair: A retrospective comparative study of proximal TIP, Onlay, and Duckett. J Pediatr Urol. 2016 Aug;12(4):198.e1-6. doi: 10.1016/j.jpurol.2016.04.034. Epub 2016 Jun 2. PMID 27318548
- [Result] Spinoit AF, Poelaert F, Van Praet C, Groen LA, Van Laecke E, Hoebeke P. Grade of hypospadias is the only factor predicting for re-intervention after primary hypospadias repair: a multivariate analysis from a cohort of 474 patients. J Pediatr Urol. 2015 Apr;11(2):70.e1-6. doi: 10.1016/j.jpurol.2014.11.014. Epub 2015 Feb 26. PMID 25797860